CLINICAL TRIAL: NCT04214444
Title: Evaluation of Prime-boost Anti-pneumococcal Vaccination in Patients With Diffuse Large B Cell Lymphoma Treated With Rituximab (EVAPOR Study)
Brief Title: Evaluation of Prime-boost Anti-pneumococcal Vaccination in Patients With Diffuse Large B Cell Lymphoma Treated With Rituximab
Acronym: EVAPOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Hôpital Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR190111-EVAPOR; 2019-002542-20 (EudraCT Number)
Record Dates: First submitted 2019-12-24; First posted 2020-01-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pneumococcal Infections; Lymphoma, Large B-Cell, Diffuse
Keywords: Lymphoma; pneumococcal vaccination; prime-boost; rituximab
MeSH Terms: conditions — Pneumococcal Infections; Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-dose before treatment (Active Comparator): 12 patients will receive a single-dose of prevenar before immunochemotherapy (R-CHOP) following two months later by pneumovax injection
  Interventions: Biological: Anti-pneumococcal vaccination with prime-boost strategy in patients with diffuse large B cell lymphoma
- Single-dose after treatment (Active Comparator): 12 patients will receive a singe-dose of prevenar three weeks after the beginning of the immunochemotherapy (R-CHOP) following two months later by pneumovax injection
  Interventions: Biological: Anti-pneumococcal vaccination with prime-boost strategy in patients with diffuse large B cell lymphoma
- Double-dose before treatment (Experimental): 12 patients will receive a double-dose of prevenar before immunochemotherapy (R-CHOP) following two months later by pneumovax injection.
  Interventions: Biological: Anti-pneumococcal vaccination with prime-boost strategy in patients with diffuse large B cell lymphoma

INTERVENTIONS:
Biological: Anti-pneumococcal vaccination with prime-boost strategy in patients with diffuse large B cell lymphoma — The investigators aim to describe efficiency and tolerability of prime-boost vaccination against pneumococcus in patients with Diffuse large B-cell Lymphoma. The investigators search to evaluate immunogenicity of prime-boost depending on the time of prevenar administration (before or after immunochemotherapy) and on the dose (single or double dose).

SUMMARY:
Pneumococcal infections remain frequent and potentially fatal. To prevent them, two anti-pneumococcal vaccines exist: a 13-valent conjugate vaccine (Prevenar®) and a 23-valent polysaccharide vaccine (Pneumovax®). For their utilization, several studies approved a prime-boost strategy. It consist two administer Pneumovax® at least two months later than Prevenar®. Patients with diffuse large B-cell Lymphoma (DLBCL) have a higher-risk to develop a pneumococcal infection. The main reason is immunosuppression, induced by rituximab (B cell depletion), chemotherapy and lymphoma. Patients are treated by immunochemotherapy, combining rituximab (anti-CD20 monoclonal antibody) and conventional chemotherapy (CHOP). However, those patients have a low rate of vaccination (about 15%).

DETAILED DESCRIPTION:
Pneumococcal infections remain frequent and potentially fatal. To prevent them, two anti-pneumococcal vaccines exist: a 13-valent conjugate vaccine (Prevenar®) and a 23-valent polysaccharide vaccine (Pneumovax®). For their utilization, several studies approved a prime-boost strategy. It consist two administer Pneumovax® at least two months later than Prevenar®. Patients with diffuse large B-cell Lymphoma (DLBCL) have a higher-risk to develop a pneumococcal infection. The main reason is immunosuppression, induced by rituximab (B cell depletion), chemotherapy and lymphoma. Patients are treated by immunochemotherapy, combining rituximab (anti-CD20 monoclonal antibody) and conventional chemotherapy (CHOP). However, those patients have a low rate of vaccination (about 15%). Also, in the current literature, rare studies investigated prime-boost immunogenicity in this relevant population. The investigators will evaluate vaccinal response of 10 serotype-specific immunoglobulin G (1, 3, 4, 6B, 7F, 9V, 14, 18C, 19F, 23F) at different time of treatment.

The investigators search to compare efficiency of prime-boost anti-pneumococcal vaccination according to the time of prevenar administration (before or after immunochemotherapy) and to the dose of Prevenar® (single or double-dose).

ELIGIBILITY:
Inclusion Criteria:

* De novo Diffuse Large B-Cell Lymphoma diagnostic (according 2016 World Health Organization (WHO) classification)
* Treatment decision by immunochemotherapy (R-CHOP)
* Age over 18 years old
* Negative pregnancy test at inclusion
* Active contraception at inclusion
* Free and informed consent procedure at inclusion
* Affiliation of the social security system

Exclusion Criteria:

* Patient with prior treatment by immunotherapy or chemotherapy
* Patient with prior treatment by debulking chemotherapy (COP)
* Patient with prior treatment by high-dose of corticosteroids
* Patients with an autoimmune disease
* Patients with a diffuse large B-cell lymphoma from transformation (follicular lymphoma, chronic lymphoid leukemia)
* Immunosuppressed patient with : asplenia, hereditary immunodeficiency disorder, infection by HIV, hepatitis B or C viruses, transplanted patient, hematopoietic stem cell transplantation, nephrotic syndrome, meningeal breach, cochlear implants.
* Patients vaccinated in the last month before inclusion
* Patients with prior transfusion of blood-products or immunoglobulins in the last three months before inclusion
* Patient with bleeding disorders or thrombopenia contraindicating intramuscular injection
* Patient with prior pneumococcal documented infection
* Patient with current pregnancy and/or breastfeeding
* Patient under curatorship or guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Proportion of responder patients at the end of treatment. | - day of Prevenar® administration, - day of Pneumovax® injection (2 months after Prevenar® injection) - six weeks after Pneumovax® injection - 1 month after last R-CHOP cycle, - at six months after end of treatment.
  The response to a specific serotype was defined as both a 2-fold increase of pneumococcal IgG antibody level (ELISA) between baseline and end of treatment (one month after last RCHOP cycle) and an antibody level >= 1µg/mL. at end of treatment.

SECONDARY OUTCOMES:
Rates of responders patients to each serotype as assessed by opsonophagocytosis | - day of Prevenar® administration, - day of Pneumovax® injection (2 months after Prevenar® injection) - six weeks after Pneumovax® injection - 1 month after last R-CHOP cycle, - at six months after end of treatment.
  response to a specific serotype was defined by both at least a fourfold increase of the opsonization index (OI, defined by the serum dilution killing 50% of the bacterial inoculum) between baseline and end of treatment.
Tolerance of the double-dose compared to single dose of Prevenar® | During the two weeks after both vaccines injection
  Presence of local and/or systemic reaction detailed on a questionary (fever, headache, fatigue, chills, rash, muscle pain, joint pain)
Clinical efficiency | During all the study (one year for each patient)
  Pneumococcal documented infection during treatment (pneumonia, meningitis, acute media otitis, bacteremia) with proof of pneumococcal presence (on blood cultures, chest radiography, other samples)

CONTACTS AND LOCATIONS:
Overall Officials: ZOHA MAAKAROUN-VERMESSE, MD-PHD, Study Director — University Hospital of TOURS
Locations (1):
- GYAN, Tours, France